CLINICAL TRIAL: NCT04425889
Title: Prevalence of SARS-CoV-2 Antibodies Among Healthcare Workers in a COVID-19 Unit
Brief Title: COVID-19 Antibodies Among Healthcare Workers
Status: Completed | Type: Observational
Sponsor: Hospital Universitario Dr. Jose E. Gonzalez (Other)
Responsible Party: Principal Investigator, Dr. Adrian Camacho-Ortiz, Head of infectious diseases, Hospital Universitario Dr. Jose E. Gonzalez
Other Study IDs: IF20-00008
Record Dates: First submitted 2020-06-06; First posted 2020-06-11 (Actual); Last update posted 2020-06-12 (Actual); Status verified 2020-06

CONDITIONS: COVID-19; SARS-CoV 2
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- exposed Healthcare workers: Healthcare workers working for 8 weeks in a COVID-19 area
  Interventions: Diagnostic Test: COVID-19 IgG/IgM Rapid Test Cassette test (Healgen Scientific, Houston, Texas, USA)

INTERVENTIONS:
Diagnostic Test: COVID-19 IgG/IgM Rapid Test Cassette test (Healgen Scientific, Houston, Texas, USA) — a blood sample is drained for detection of IgG and IgM antibody

SUMMARY:
Observational, point of prevalence study determining the presence of anti-SARS-CoV-2 antibody

DETAILED DESCRIPTION:
All Healthcare workers (HCW) who had entered contaminated areas at least once and that 14 days or more had passed from their first entrance to contaminated areas were included. They were classified as asymptomatic and pauci-symptomatic. A COVID-19 IgG/IgM rapid test was used for antibody detection, and selected participants were subject to real time polymerase chain reaction (qPCR) for SARS-CoV-2.

ELIGIBILITY:
Inclusion Criteria:

* All healthcare workers who had entered contaminated areas at least once and that 14 days or more had passed from their first entrance were included

Exclusion Criteria:

* Healthcare workers who did not have exposure for more or equal 14 days
* Healthcare workers who did not wish to participate

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthcare workes of any category that are 18 years of age or older, who work in the COVID-19 unit at the University Hospital and hve been diagnosing and treating suspected or confirmed cases of COVID-19
Sampling Method: Non-Probability Sample
Enrollment: 156 (Actual)
Dates: Start 2020-05-05 (Actual); Primary Completion 2020-05-30 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
Presence of antibody | through study completion, an average of 8 weeks
  presence of IgG and/or IgM against SARS-CoV-2

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario José E. Gonzalez, Monterrey, Nuevo León, Mexico

IPD SHARING:
Plan to Share IPD: Undecided